CLINICAL TRIAL: NCT04330729
Title: The Effect of Low-dose Salicylate Treatment on Platelet Function in Patients With Renal Failure Treated With Darbepoetin Alfa
Brief Title: The Effect of Salicylate on Platelet Function in CKD (Chronic Kidney Disease) Patients Treated With Aranesp
Acronym: EPOASA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-018-2018
Record Dates: First submitted 2020-03-20; First posted 2020-04-01 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-12

CONDITIONS: Erythropoietin Adverse Reaction
Keywords: hemodialysis; platelet function; erythropoietin; thrombosis; anaemia
MeSH Terms: conditions — Thrombosis; Anemia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dialysis patients (Experimental): Patients will tablet acetylsalicylic acid 75mg x 1 for 4 weeks.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — Se arm description

SUMMARY:
The aim of the study is to

1. To determine whether treatment with Erythropoiesis-stimulating agents (in the form of Aranesp®) affects platelet function, and how.
2. To determine whether salicylate treatment changes the effect of EPO (erythropoietin) on platelet function.

DETAILED DESCRIPTION:
Background:

It is well known that treatment with EPO increases the risk of thrombotic complications in patients with chronic kidney disease, including cerebral thrombosis. The requited level of Hgb for sufficient treatment has therefore been set at a relatively low level (6.8-7.3 mM). One obvious potential cause of this problem is the increased thrombocytosis and platelet activation caused by EPO treatment. An old investigation has shown that low-dose acetyl salicylic acid (ASA) treatment can remove this effect. This investigation has not been performed using modern methods to investigate platelet function, and the possible prophylaxis of EPO-induced thrombosis has since received little interest.

Investigators of current study therefore propose to repeat this investigation using advanced methods for assessing thrombocyte function, as a preliminary, exploratory investigation prior to a later randomized controlled study.

Pre-treatment Washout (4 weeks, 6 weeks if treated with Mircera))

Patients who are not treated with ESA do not receive any treatment. Patients treated with ESA stop their treatment for 4 weeks. Patients treated with Mircera ® stop treatment for 6 weeks.

Patients must not take ASA as an analgesic during the whole period of the project.

At the end of the pre-treatment period, the Standard package (blood samples) is assessed.

EPO Treatment (4 weeks) The patient is treated with darbepoetin alfa (Aranesp) in equipotent doses compared to previous therapy.

After 2 weeks the Hgb is measured, and the EPO dosis adjusted if necessary at the discretion of the responsible physician.

After 4 weeks, the Standard package is assessed. If the Hgb is >8,0 mM or is rising rapidly (>1,2mM per month), the EPO dose is reduced at the discretion of the responsible physician.

EPO + ASA Treatment Aranesp treatment is supplemented with ASA (Hjertemagnyl ® 75 mg x 1 daily). After 4 weeks the Standard package is assessed.

If the patient develops gastrointestinal symptoms (abdominal pain, nausea or heartburn), and is not already being treated with pantoprazole or other PPI (proton pump inhibitors), treatment is supplemented with pantoprazole 40 mg x 1 daily.

ASA treatment withdrawal - e.g. in regard to surgery - results in discontinuation of participation in the study.

Post-treatment Washout Both Aranesp and Hjertemagnyl treatment is stopped. After 4 weeks the Standard package and is assessed.

Termination The indication for, and dose of ESA and ASA is prescribed at the discretion of the responsible physician.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis, peritoneal dialysis or CKD 5 treated conservatively
* aged 18-85
* indication for treatment with Erythropoiesis-stimulating agents (ESA)

Exclusion Criteria:

1. Known allergy to ASA
2. Known contraindication to ASA, e.g. recent bleeding episode.
3. Known indication for ASA. If the patient is being treated with ASA, and the physician does not find any indication for this treatment, this can be stopped, and the patient included after 4 weeks.
4. Raised reticulocyte count
5. Current anticoagulant therapy, e.g. warfarin, ADP receptor inhibitor (excepting short-term anticoagulant therapy in connection with dialysis)
6. Short expected length of life
7. Inability to give informed consent
8. Expected non-compliance
9. Active cancer - except for non-melanoma skin-cancer
10. Iron deficiency (defined as a reticulocyte Hgb <1,8 fmol. Patients can be included when their iron deficiency has been cured. .
11. Change in ESA dosis >33,3% within previous 2 month
12. Fertile women. Pregnancy is excessively rare in dialysis patients. Women who are <50 years, or who are still menstruating will be excluded from the study.
13. Stable Aranesp ® dose <20 µg/week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Thrombocytaggregometry | 16 weeks
  Multiplate induced with arachidonic acid, ADP (adenosine diphosphate) and TRAP (Thrombin receptor-activating peptid)

SECONDARY OUTCOMES:
D-dimer | 16 weeks
  D-dimer, (FEU mg/L)
MPV | 16 weeks
  Mean platelet volume, (fL=femtoliters)
Total platelet count | 16 weeks
  Total platelet count (units per milliliters)
PDW | 16 weeks
  platelet distribution width (fL = femtoliters)
IPC | 16 weeks
  immature platelet count (platelets/microliter)
IPF | 16 weeks
  Immature platelet fraction (%)
H-IPF | 16 weeks
  Highly immature platelet fraction (%)
ROTEM | 16 weeks
  Thromboelastometry
TGF-beta | 16 weeks
  Transforming growth factor beta
sP-selectin | 16 weeks
  Soluble platelet selectin
Thrombomodulin | 16 weeks
  Thrombomodulin

CONTACTS AND LOCATIONS:
Overall Officials: James G Heaf, Study Director — Department of medicine, Zealand University Hospital, Denmark
Locations (1):
- Medicinsk afdeling, SUH Roskilde, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No